CLINICAL TRIAL: NCT07333937
Title: Neratinib Combined With Fulvestrant and Eribulin in the Treatment ofHR+/HER2+ Advanced Breast Cancer After Trastuzumab Deruxtecan Resistance:A Single-Arm, Multicenter, Exploratory Clinical Study
Brief Title: Neratinib Combined With Fulvestrant and Eribulin in the Treatment ofHR+/HER2+ Advanced Breast Cancer
Acronym: NETHER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJYY-KY-20252554
Record Dates: First submitted 2025-12-14; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Brest Cancer
Keywords: Neratinib; Fulvestrant; Eribulin; HR+/HER2+ Advanced Breast Cancer
MeSH Terms: interventions — Fulvestrant; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neratinib Combined with Fulvestrant and Eribulin (Experimental): Neratinib Combined with Fulvestrant and Eribulin after Trastuzumab Deruxtecan Resistance
  Interventions: Drug: Neratinib Combined with Fulvestrant and Eribulin

INTERVENTIONS:
Drug: Neratinib Combined with Fulvestrant and Eribulin — neratinib combined with fulvestrant and eribulin in the treatment of HR+/HER2+ advanced breast cancer after trastuzumab deruxtecan resistance

SUMMARY:
This study aims to explore the efficacy and safety of neratinib combined with fulvestrant and eribulin in the treatment of HR+/HER2+ advanced breast cancer after trastuzumab deruxtecan resistance. The treatment regimen of neratinib + fulvestrant + eribulin in this study is expected to provide a new and effective therapeutic strategy for patients with triple-positive breast cancer who develop resistance to trastuzumab deruxtecan, and offer novel therapeutic insights for advanced triple-positive breast cancer.

DETAILED DESCRIPTION:
This study is a single-arm, exploratory clinical trial. Eligible patients with recurrent or metastatic breast cancer will be screened and enrolled after signing the informed consent form, and will receive neratinib combined with fulvestrant and eribulin until disease progression or intolerable toxicity occurs. During the treatment period, clinical tumor imaging assessments will be performed every 6 weeks (2 cycles) in accordance with RECIST v1.1; safety assessments will be conducted using NCI-CTCAE 5.0, and adverse events will be recorded throughout the study and within 30 days after the end of treatment (the recording period for serious adverse events or adverse events related to the drugs involved in this trial will be extended to 90 days after the end of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years and ≤75 years;
* ECOG performance status of 0-2;
* Histologically confirmed HR-positive/HER2-positive advanced breast cancer:
* Definition of HER2 positivity: IHC 3+ or IHC 2+/ISH positive prior to T-DXd treatment;
* Definition of HR positivity: ER or PR ≥1%;
* Refractory to prior treatment containing T-DXd (definition of resistance: a. Definite disease progression per RECIST v1.1 criteria; b. Intolerance to T-DXd treatment);
* Prior exposure to anthracyclines and taxanes (including use in the adjuvant/neoadjuvant setting);
* Presence of at least one measurable lesion (per RECIST v1.1 criteria);
* Estimated survival time ≥3 months;
* Adequate function of major organs, meeting the following requirements (no blood transfusion, no use of leukocyte- or platelet-stimulating agents within 2 weeks prior to screening);
* For premenopausal or non-surgically sterilized female patients: Agreement to abstain from sexual activity or use effective contraceptive methods during treatment and for at least 7 months after the last dose of study treatment;
* Voluntary participation in the study, signing of the informed consent form, good compliance, and willingness to cooperate with follow-up.

Exclusion Criteria:

* Severe allergic reactions to neratinib, eribulin, fulvestrant, or any of their excipients;
* Prior treatment with neratinib, other small-molecule anti-HER2 TKIs, or eribulin;
* Patients with inflammatory breast cancer;
* A history of other malignant tumors within the past 5 years or concurrent malignant tumors (including cured malignant tumors such as carcinoma in situ of the cervix, basal cell carcinoma, or squamous cell carcinoma);
* Concurrent receipt of anti-tumor therapies in other clinical trials, including endocrine therapy, bisphosphonate therapy, or immunotherapy;
* Receipt of major surgical procedures unrelated to breast cancer within 4 weeks prior to enrollment, or failure to fully recover from such surgical procedures;
* Severe cardiac diseases or disorders, including but not limited to: --Documented history of heart failure or systolic dysfunction (LVEF < 50%); --High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate > 100 bpm, significant ventricular arrhythmias (e.g., ventricular tachycardia), or high-grade atrioventricular block (i.e., Mobitz II second-degree atrioventricular block or third-degree atrioventricular block);
* Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg);
* Inability to swallow, intestinal obstruction, or other factors affecting drug administration and absorption;
* Known history of allergies to any components of the study drugs; history of immunodeficiency (including positive HIV test results), other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
* Pregnant or lactating female patients; female patients of childbearing potential with a positive baseline pregnancy test; or fertile patients unwilling to use effective contraceptive methods throughout the trial and for 7 months after the last dose of study treatment;
* Severe comorbid diseases or other concurrent conditions that may interfere with the planned treatment, or any other circumstances deemed by the investigator to make the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-11-20 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From treatment initiation to disease progression, intolerable toxicity, or study completion, whichever occurs first，assessed up to 10 months
  The proportion of patients whose tumor lesions achieve "Partial Response (PR)" or "Complete Response (CR)" after treatment

SECONDARY OUTCOMES:
progression free survival | From first treatment initiation to the first occurrence of disease progression (per RECIST v1.1) or death from any cause, or study completion (whichever occurs first)，assessed up to 60 months
  the length of time from a patient's enrollment to the first occurrence of either "disease progression (PD)" or "death from any cause".
overall survival | From first treatment initiation to death from any cause or study completion, whichever occurs first, with a minimum follow-up of 12 months for surviving patients，assessed up to 100 months
  the length of time from a patient's enrollment to death from any cause
Disease control rate | From first treatment initiation to disease progression, intolerable toxicity, or study completion (whichever occurs first), with disease control status confirmed for ≥4 weeks per RECIST v1.1
duration of response | From the first confirmed Complete Response (CR) or Partial Response (PR) (per RECIST v1.1, maintained for ≥4 weeks) to the first documented disease progression (PD) or death from any cause, or study completion，assessed up to 10 months
adverse effects | From the first dose of study treatment (neratinib + fulvestrant + eribulin) to 30 days after the last dose of study treatment. For serious adverse events (SAEs), the follow-up and recording period is extended to 90 days after the last dose.

IPD SHARING:
Plan to Share IPD: No